CLINICAL TRIAL: NCT03218202
Title: Stricture Definition and Treatment (STRIDENT) Observational Study.
Acronym: STRIDENT
Status: Terminated | Type: Observational
Why Stopped: To focus on STRIDENT intervention studies as this study population is heterogenous
Sponsor: St Vincent's Hospital Melbourne (Other)
Collaborators: Australasian Gastro Intestinal Research Foundation (Other)
Responsible Party: Principal Investigator, Michael Kamm, Professor of Gastroenterology, St Vincent's Hospital Melbourne
Other Study IDs: SVHMelbourneSTRIDENT3
Record Dates: First submitted 2017-07-07; First posted 2017-07-14 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis; Stricture; Colon
Keywords: Inflammatory Bowel Disease; Crohn Disease; Ulcerative Colitis; Intestinal stricture
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Constriction, Pathologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Standard blood tests. Tests for Single Nucleotide Polymorphisms. Stool testing, Tissue Sampling.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Two thirds of patients with Crohn's disease require intestinal surgery at some time in their life. Intestinal strictures, that is narrowing of the bowel due to inflammation and scarring, are the most common reason for surgery. Despite the high frequency, associated disability, and cost there are no are no treatment strategies that aim to improve the outcome of this disease complication. The STRIDENT (stricture definition and treatment) studies aim to determine biochemical and imaging features associated with the development of strictures and in related STRIDENT studies develop strategies for treatment.

DETAILED DESCRIPTION:
Patients with asymptomatic Crohn's disease strictures will be followed prospectively for 12 months using imaging (including MRI/intestinal ultrasound) and biochemical analyses (including CRP/calprotectin). Patient's with symptomatic or asymptomatic ulcerative colitis related strictures will be followed similarly. Risk factors for progression of strictures and development of symptoms will be identified.

ELIGIBILITY:
Inclusion Criteria:

* Inflammatory bowel disease patients with intestinal stricture(s) identified on CT, MRI or endoscopy but without associated symptoms

Exclusion Criteria:

* Low rectal or anal strictures
* Evidence of dysplasia or malignancy from stricture biopsies or adjacent mucosal biopsies
* Patients for whom endoscopy is not suitable due to co-morbidities or clinical state
* Inability to give informed consent
* Suspected perforation of the gastrointestinal tract
* Inability to undergo MRI small bowel due to a contraindication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with inflammatory bowel disease (Crohn's Disease or Ulcerative Colitis) without symptoms who are incidentally found to have a stricture on CT, MRI or endoscopy.
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-08-29 (Actual)

PRIMARY OUTCOMES:
Development of symptoms | 12 months
  Number of patients who develop symptoms and require step up in therapy (drug, endoscopic or surgical therapy).

SECONDARY OUTCOMES:
Imaging features associated with development of symptoms (MRI). | 12 months
  MaRIA
Imaging features associated with development of symptoms (Intestinal Ultrasound). | 12 months
  Limberg's score
Biochemical features associated with development of symptoms | 12 months
  CRP and calprotectin
Patient reported outcomes | 12 months
  SF36
Patient reported outcomes | 12 months
  IBDQ
Requirement for step up in drug therapy | 12 months
  Need for additional drug therapy due to development of symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Emily Wright, MBBS PhD, Principal Investigator — St Vincent's Hospital Melbourne; Bronte Holt, MBBS PhD, Principal Investigator — St Vincent's Hospital Melbourne; Michael Kamm, MBBS PhD, Principal Investigator — St Vincent's Hospital Melbourne
Locations (1):
- St. Vincent's Hospital Melbourne, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided